CLINICAL TRIAL: NCT06637423
Title: A Phase 1/2 Open-label Clinical Study to Evaluate the Safety and Efficacy of Intravesical Sacituzumab Tirumotecan (Sac-TMT, MK-2870) in Participants With Intermediate-risk Non-muscle Invasive Bladder Cancer (NMIBC)
Brief Title: A Clinical Study of Sacituzumab Tirumotecan (MK-2870) in Patients With Bladder Cancer (MK-2870-027)
Acronym: TroFuse-027
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2870-027; 2024-514983-23-00 (Registry Identifier: EU CT); U1111-1308-6998 (Registry Identifier: UTN); MK-2870-027 (Other: MSD)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-Muscle Invasive Bladder Cancer
Keywords: Non-Muscle Invasive Bladder Cancer; Low Grade; Intermediate Risk; Recurrent Low-Grade
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sacituzumab tirumotecan (Experimental): Participants receive intravesical Sacituzumab Tirumotecan for 6 weeks
  Interventions: Drug: Sacituzumab tirumotecan; Drug: Rescue medication; Drug: Supportive care measures

INTERVENTIONS:
Drug: Sacituzumab tirumotecan — Intravesical administration
  Other Names: SKB264; sac-TMT; MK-2870
Drug: Rescue medication — Participants are allowed to take rescue medication for stomatitis or oral mucositis. At the discretion of the investigator, participants are provided with a prescription for rescue medications. Recommended rescue medications are antihistamine, histamine-2 (H2) receptor antagonist, acetaminophen or equivalent, dexamethasone or equivalent infusion or steroid mouthwash (dexamethasone or equivalent), antiemetic medications, oral nystatin suspension or antifungal medications, antidiarrheal agents, antiemetic agents, opiate and non-opiate analgesic agents, appetite stimulants, and granulocyte and erythroid growth factors.
Drug: Supportive care measures — Participants are allowed to take supportive care measures for the management of adverse events associated with study intervention at the discretion of the investigator. Artificial tear drops or gel may be given as a supportive care for Ocular Surface Toxicity.

SUMMARY:
The goal of the study is to learn about the safety of Sacituzumab Tirumotecan and if people can tolerate it when given in the bladder and find the highest dose that people can take without having certain problems. Researchers will then choose a dose level of Sacituzumab Tirumotecan to use in future studies to learn how well the drug works.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Has recurrent low-grade (Ta) Non-Muscle Invasive Bladder Cancer (NMIBC) in the bladder
* Must have visible tumor by cystoscopy within 12 weeks prior to first dose
* Has intermediate-risk NMIBC defined as 1 or more of the following risk factors:

  * Multiple tumors
  * >1 occurrence of low-grade NMIBC within 1 year of the current diagnosis at Screening
  * Early recurrence (<1 year) of the initial diagnosis of low-grade disease
  * Solitary tumor >3 cm
  * Failure of prior intravesical treatment
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 assessed within 14 days prior to first dose

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Newly diagnosed low-grade non-muscle invasive bladder cancer (Ta NMIBC) in the bladder
* Past or current history of high-grade (Ta or T1 or CIS) NMIBC, muscle invasive bladder cancer (MIBC) or metastatic urothelial carcinoma (UC)
* Has a condition that would prohibit normal voiding (or hold bladder voiding for 1 to 2 hours)
* Has history of documented severe dry eye syndrome, severe Meibomian gland disease, and/or blepharitis, or severe corneal disease that prevents and/or delays corneal healing
* Has active inflammatory bowel disease requiring immunosuppressive medication or previous history of inflammatory bowel disease (eg, Chron's disease, ulcerative colitis, or chronic diarrhea)
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease
* Known additional malignancy that is progressing or has required active treatment within the past 3 years
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity (DLT) | Up to approximately 7 weeks
  DLT will be defined as any drug-related adverse event (AE) observed during the DLT evaluation period (7 weeks). All toxicities will be graded using National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) version 5.0.
Number of Participants Experiencing an Adverse Event (AE) | Up to approximately 10 weeks
  An AE is defined as any untoward medical occurrence in a participant administered a study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of participants who experience an AE will be reported.
Number of Participants Discontinuing Study Treatment due to an Adverse Event (AE) | Up to approximately 6 weeks
  An AE is defined as any untoward medical occurrence in a participant administered a study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of participants who discontinue study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Area Under the Serum Concentration-Time Curve (AUC) of sacituzumab tirumotecan (sac-TMT) Antibody-Drug Conjugate (ADC) | Up to approximately 6 weeks
  Blood samples will be collected to determine the AUC of sac-TIMT ADC
Maximum Serum Concentration (Cmax) of sac-TMT ADC | Up to approximately 6 weeks
  Blood samples will be collected to determine the Cmax of sac-TMT ADC
Minimum Serum Concentration (Cmin) of sac-TMT ADC | Up to approximately 6 weeks
  Blood samples will be collected to determine the Cmin of sac-TMT ADC
Serum Apparent terminal half-life (t½) of sac-TMT ADC | Up to approximately 6 weeks
  Blood samples will be collected to determine the t1/2 of sac-TMT ADC
Serum AUC of sac-TMT Total Antibody (TAb) | Up to approximately 6 weeks
  Blood samples will be collected to determine the AUC of sac-TMT Tab
Serum Cmax of sac-TMT Tab | Up to approximately 6 weeks
  Blood samples will be collected to determine the Cmax of sac-TMT Tab
Serum Cmin of sac-TMT Tab | Up to approximately 6 weeks
  Blood samples will be collected to determine the Cmin of sac-TMT Tab
Serum t½ of sac-TMT Tab | Up to approximately 6 weeks
  Blood samples will be collected to determine the t1/2 of sac-TMT Tab
Plasma AUC of sac-TMT payload | Up to approximately 6 weeks
  Blood samples will be collected to determine the AUC of sac-TMT payload
Plasma Cmax of sac-TMT payload | Up to approximately 6 weeks
  Blood samples will be collected to determine the Cmax of sac-TMT payload
Plasma Cmin of sac-TMT payload | Up to approximately 6 weeks
  Blood samples will be collected to determine the Cmin of sac-TMT payload
Plasma t½ of sac-TMT payload | Up to approximately 6 weeks
  Blood samples will be collected to determine the t1/2 of sac-TMT payload
Complete Response Rate (CRR) | Up to approximately 6 months
  CRR is defined as the percentage of participants who will be absent of residual tumor in the bladder assessed locally by cystoscopy evaluation and negative urine cytology and/or biopsy and imaging if applicable.
Duration of Complete Response (DCR) | Up to approximately 24 months
  Duration of CR for participants who demonstrate CR is defined as the time from the first documented evidence of CR (absence of residual tumor in the bladder assessed locally by cystoscopy evaluation and negative urine cytology and/or biopsy and imaging if applicable) until the occurrence of histologically confirmed nonmuscle invasive urothelial carcinoma (UC) by local pathology review or locally advanced or metastatic UC, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (13):
- United States (4):
  - Michael G Oefelein Clinical Trials ( Site 0053), Bakersfield, California
  - Moffitt Cancer Center ( Site 0057), Tampa, Florida
  - Northwestern University ( Site 0051), Chicago, Illinois
  - Johns Hopkins University ( Site 0055), Baltimore, Maryland
- Canada (2):
  - Princess Margaret Cancer Centre ( Site 0003), Toronto, Ontario
  - CIUSSS de l'Estrie-CHUS ( Site 0002), Sherbrooke, Quebec
- France (3):
  - Hôpital Claude Huriez ( Site 0012), Lille, Nord
  - HENRI MONDOR HOSPITAL ( Site 0011), Créteil, Val-de-Marne
  - Gustave Roussy ( Site 0013), Villejuif, Val-de-Marne
- Erasmus Medisch Centrum ( Site 0032), Rotterdam, South Holland, Netherlands
- Spain (2):
  - Hospital Universitario Virgen de la Victoria ( Site 0043), Málaga, Andalusia
  - Hospital Universitario 12 de Octubre ( Site 0042), Madrid
- St Bartholomew s Hospital ( Site 0061), London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/